CLINICAL TRIAL: NCT04270019
Title: The Use of Polyethylene Glycol to Improve Sensation Following Digital Nerve Laceration: A Randomized Controlled Trial
Brief Title: Polyethylene Glycol to Improve Sensation Following Digital Nerve Laceration
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of staff, REB closed the file due to expired renewal
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0644
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Nerve Injury; Nerve Injury
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — polyethylene glycol 3350; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, double-blind, placebo-controlled human clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): This group will receive polyethylene glycol (50% weight/volume) applied to the nerve coaptation site during primary repair of peripheral nerve injury in the hand.
  Interventions: Drug: Polyethylene Glycol 3350
- Control (Placebo Comparator): This group will receive normal saline applied to the nerve coaptation site during primary repair of peripheral nerve injury in the hand.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — In order to prepare PEG 3350 50% weight/volume, 25 grams of the sterilized PEG 3350 will be measured out and placed into a sterilized glass bottle then 25 mL of sterile water will be added. The solution will be allowed to rest for 10 minutes so that dissolution may occur. More sterile water will then be added so the total volume is 50mL. This solution will then be sterilized by the Halifax Health Infirmary pharmacy department using a liquid autoclave cycle of 120 degrees Celsius for 20 minutes in a glass vial. The 50 mL solution will be portioned into 2mL sterilized glass vials using a standard aseptic technique. The solutions will be kept at a solid frozen state between negative 25 degrees Celsius and negative 10 degrees Celsius for a maximum of 45 days. The solutions will be removed from storage on the day of surgical utilization in order to ensure storage guidelines are kept to the highest standards.
  Arms: Experimental
Drug: Normal Saline — Standard solution of sterile normal saline.
  Arms: Control

SUMMARY:
PEG is a fusogen, a type of chemical that aids in mediating cell fusion. PEG helps nerve cells recover neuronal continuity by removing plasmalemmal-bound water which opens the axonal ends on both sides of the injury. Opening axonal ends permits the nerve ends to reconnect and begin regeneration. PEG has been tested on animal models extensively and in earthworm models has been shown to induce fusion rates in 80-100% of neuronal cells. In crushed or severed mammalian sciatic nerves PEG has enhanced neuronal continuity to baseline functioning levels.

Human applications for PEG have been tested by Bamba and colleagues in a case series with encouraging results. No studies, to our knowledge, have prospectively examined the use of PEG in peripheral nerve injuries. We propose a placebo controlled, double-blinded randomized controlled trial to test the hypothesis that local PEG administration can enhance sensory nerve regeneration following digital nerve transection compared to surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* (1) surgery within twenty-four hours of injury (2) surgery completed in the minor procedures unit of the Halifax Infirmary.

Exclusion Criteria:

* (1) patients with cognitive impairment

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Sensory Recovery | Testing to be done at one month, three months, and six months post-operatively.
  Sensory recovery will be assessed by a blinded and trained OT through standardized testing with static two point discrimination (s2PD) and Semmes-Weinstein monofilament testing (SWMT). The end point will be composite in nature as both s2PD and SWMT are important to gauge and are the gold standards in determining sensory recovery.

SECONDARY OUTCOMES:
Functional Recovery | Administered six months post-operatively. Maximum score of 100, minimum score of 0. A higher score means better functional recovery.
  Functional recovery assessed by the Michigan Health Questionnaire (MHQ).

IPD SHARING:
Plan to Share IPD: No